CLINICAL TRIAL: NCT05645081
Title: PREDICT-EV; the Association of Extracellular Vesicles and Dysregulated Coagulation in the Prediction of Stroke
Brief Title: Extracellular Vesicles and Dysregulated Coagulation in the Prediction of Stroke
Acronym: PREDICT-EV
Status: Recruiting | Type: Observational
Sponsor: Cwm Taf University Health Board (NHS) (Other Government)
Collaborators: Cardiff Metropolitan University (Other)
Responsible Party: Sponsor
Other Study IDs: CT/1245/281530/19/20
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-02

CONDITIONS: Stroke, Ischemic; Transient Ischemic Attack; Coagulation Disorder
Keywords: Stroke Risk; Transient Ischemic Attack; Extracellular Vesicles; Pro-Thrombotic Risk
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy Control: A group of participants with no previous symptoms or diagnosis of TIA or stroke.
- Non-TIA Control: A group of participants who were referred to TIA clinic with symptoms of a TIA, however, were subsequently confirmed as not suffering with a TIA.
- TIA, non-stroke: A group of participants who were confirmed as suffering a TIA by a stroke clinician following admission to hospital, admission to Accident and Emergency or after being referred to TIA clinic. These participants did not suffer a stroke within 12 months of TIA diagnosis.
- TIA, stroke: A group of participants who were confirmed as suffering a TIA by a stroke clinician following admission to hospital, admission to Accident and Emergency or after being referred to TIA clinic. These participants went on to suffer a stroke within 12 months of TIA diagnosis.

SUMMARY:
Annually 100,000 strokes occur, placing stroke as the largest cause of disability in the UK. 90% of strokes are preventable, leading to national focus on programmes including "The National Stroke Programme" to act on preventing, treating, and improving post-stroke care. Importantly, over 25% of ischaemic stroke sufferers have previously had a Transient Ischaemic Attack (TIA), which presents the biggest concern for TIA patients. There are no measures which reliably identify TIA patients most likely to suffer a stroke. Novel biomarkers for predicting stroke are key to addressing this problem. The PREDICT-EV study aims to screen 300 TIA patients and follow them over 12-months. The investigators will determine if a novel biomarker we've identified to increase thrombotic risk (endothelial derived extracellular vesicles) and the resulting increased prothrombin time is associated with patients at highest risk of stroke.

ELIGIBILITY:
The inclusion criteria for phase 1 (initial patient recruitment) will be:

1. Patients with or without diagnosis of TIA made by a physician working in stroke medicine, sufficiently so to start post-TIA care or so that no further investigation is thought necessary to confirm or refute the diagnosis.
2. TIA confirmed patient has been prescribed antiplatelet drugs or anticoagulants.
3. Patients must be aged > 18 years.
4. Patients are taking an ordinary diet by mouth.

The inclusion criteria for phase 2 (patient representing with stroke) will be:

1. Radiological evidence, on CT and/or MR imaging of the brain of cerebral infarction, with or without secondary haemorrhage.
2. The underlying mechanism of cerebral infarction is embolic from a cardiac source (e.g. atrial fibrillation), atherothromboembolic (from aorta or other large vessels in the neck) or in-situ thrombosis. No further investigations are thought necessary to confirm or refute the diagnosis.
3. No further investigations are thought necessary to confirm or refute the diagnosis.
4. Patients must be aged >18 years.
5. Patients must not be pregnant or breast feeding.
6. Patients are taking an ordinary diet by mouth. Exclusion Criteria

The Exclusion criteria for phase 1 (initial patient recruitment) will be:

1. Inability to give consent.
2. Inability to feed by mouth.
3. Short life expectancy.
4. Pregnancy or breastfeeding.
5. Symptoms are readily explained by medical problems not involving focal cerebral ischaemia.

The Exclusion criteria for phase 2 (patient representing with stroke) will be:

1. Patients who have not previously given consent for follow up blood sampling.
2. Patients who are unable to feed by mouth.
3. Patients in whom life expectancy is short.
4. Patient is pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample will be selected from patients attending TIA clinic appointments, following primary care referral. Participants may also be identified from accident and emergency or following admission into hospital.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in the endothelial derived extracellular vesicle population | 3 years
Change in patient Prothrombin time | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Charles Hospital, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: No